CLINICAL TRIAL: NCT05075070
Title: Immunogenicity and Safety of an Inactivated COVID-19 Vaccine in People With Human Immunodeficiency Virus Infected
Brief Title: Immunogenicity and Safety of an Inactivated COVID-19 Vaccine in People With HIV Infected
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Zhejiang Provincial Center for Disease Control and Prevention (Other Government); Beijing Institute of Biological Products Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BIBP2021HIV
Record Dates: First submitted 2021-10-05; First posted 2021-10-12 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; HIV Infections
MeSH Terms: conditions — COVID-19; HIV Infections

STUDY DESIGN:
Intervention Model Description: subjects infected with HIV receive two doses inactivated COVID-19 vaccine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): A total 400 HIV-infected subjects receive two doses inactivated COVID-19 vaccine with the interval of 21 days.
  Interventions: Biological: Inactivated COVID-19 vaccine

INTERVENTIONS:
Biological: Inactivated COVID-19 vaccine — two doses inactivated COVID-19 vaccine

SUMMARY:
Evaluation of immunogenicity and safety of the subjects infected with HIV to receive the schedule of two doses inactivated COVID-19 vaccine with the interval of 21 days .

DETAILED DESCRIPTION:
The subjects infected with HIV were recruited to receive the schedule of two doses inactivated COVID-19 vaccine with the interval of 21 days .

Blood samples will be collected 2 times: before the 1st dose of vaccinatioin and 28 days after the 2nd dose of vaccination.

Any local or systemic adverse events that occurred within 21 days after vaccination will be recorded.

ELIGIBILITY:
Inclusion criteria:

* Subjects aged ≥18.
* Body temperature < 37.3 ° C confirmed by clinical examination before enrollment .
* CD4+ count is less than 500/ul and more than 50/ul .
* Female subjects of reproductive age declare that they are not pregnant, have no birth plan in the first 3 months after enrollment, and have taken effective contraceptive measures in the first 2 weeks before enrollment.
* Able and willing to complete the entire study plan during the study follow-up period.
* Have the ability to understand the study procedures, voluntarily sign informed consent, and comply with the requirements of the clinical study protocol.

Exclusion criteria for the first dose:

* Being allergic to any component of vaccines (including excipients) .
* Subjects who have experienced severe allergic reactions to vaccines (e.g. acute anaphylaxis, urticaria, angoneeurotic edema, dyspnea, etc.).
* Having uncontrolled epilepsy and other progressive neurological disorders and a history of Guillain-Barre syndrome.
* Pregnant and lactating women.
* The subjects are suffering from an acute illness; Or thrombocytopenia patients with platelet count < 20×10^9/L within three days before inoculation, that is, patients at high risk of spontaneous bleeding.
* Acute HIV infection and opportunistic infection.
* Subjects with co-opportunistic infections who did not receive antiviral therapy.
* Subjects with CD4+ count less than 50/ul who have not received antiviral therapy.
* HIV-infected subjects undergoing treatment with severe drug interactions and overlapping toxicity (kidney damage, liver damage, hematological problems, etc.).
* Patients with malignant tumors are undergoing chemotherapy and radiotherapy before and after surgery.
* Other subjects whose physical conditions, as determined by the investigator, are not suitable for inclusion in clinical studies.

Exclusion criteria for the second dose:

* Subjects who had vaccine-related adverse reactions after the first dose.
* Having high fever (axillary temperature ≥39.0℃) for three days after the first dose of inoculation, or severe allergic reaction.
* Having any adverse nervous system reaction after the first dose.
* During the acute onset of a chronic disease, or the recovery of acute complications less than two weeks.
* Subjects with severe immunodeficiency (CD4+ count less than 50/ul).
* Acute HIV infection and opportunistic infection.
* Subjects with co-opportunistic infections who did not receive antiviral therapy.
* HIV-infected subjects undergoing treatment with severe drug interactions and overlapping toxicity (kidney damage, liver damage, hematological problems, etc.).
* Other reasons for exclusion considered by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate | 28 days after the 2th dose (Day 49)
  The rate of seroconversion against coronavirus
Baseline neutralizing antibody level | Before vaccination (Day 0)
  Neutralizing antibody geometric mean titer(GMT) against coronavirus before vaccination
Neutralizing antibody level | 28 days after the 2th dose(Day 49)
  Neutralizing antibody GMT against coronavirus after the 2th dose

SECONDARY OUTCOMES:
Adverse events rate | 0-21days following vaccinations
  Analyse the incidence of adverse events following vaccination, both solicited and unsolicited
Serious adverse event rate | 0-6 months
  Report and analyse serious adverse events
Baseline T cell count | before vaccination (Day 0)
  T cell count （CD4+T，CD8+T，etc.）
Baseline HIV viral load | before vaccination (Day 0)
  HIV viral load
T cell count | 28 days after the 2th dose (Day 49)
  T cell count （CD4+T，CD8+T，etc.）
HIV viral load | 28 days after the 2th dose (Day 49)
  HIV viral load

CONTACTS AND LOCATIONS:
Overall Officials: Hanqing He, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Zhejiang provincial center for disease control and prevention, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Deng X, Dai R, Fu J, Ding L, Hu X, Sun P, Shu R, Chen L, Xu X. Inadequate immune response to inactivated COVID-19 vaccine among older people living with HIV: a prospective cohort study. J Virol. 2025 Sep 23;99(9):e0068825. doi: 10.1128/jvi.00688-25. Epub 2025 Aug 21. PMID 40838719
- [Derived] Wang Y, Li J, Zhang W, Liu S, Miao L, Li Z, Fu A, Bao J, Huang L, Zheng L, Li E, Zhang Y, Yu J. Extending the dosing interval of COVID-19 vaccination leads to higher rates of seroconversion in people living with HIV. Front Immunol. 2023 Mar 2;14:1152695. doi: 10.3389/fimmu.2023.1152695. eCollection 2023. PMID 36936952